CLINICAL TRIAL: NCT06766604
Title: Exploratory In-vitro Study Evaluating the Addition of Super-GDF9 During Capacitation-in-vitro Maturation (CAPA-IVM) of Donated Human Cumulus-oocyte Complexes (COCs) Derived From Small Antral Follicles
Brief Title: Effect of Super-GDF9 on CAPA-IVM of COCs From Small Antral Follicles
Acronym: sGDF-9
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/24/DD-BVMD
Record Dates: First submitted 2024-12-24; First posted 2025-01-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: In Vitro Fertilization
Keywords: CAPA-IVM; super-GDF9; Culture; OSFs; PCOS

STUDY DESIGN:
Intervention Model Description: Sibling oocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super-GDF9 supplementation during CAPA-IVM (Experimental): Group 1: donated COCs will be cultured in the CAPA step and the IVM step, with the addition of Super-GDF9 during CAPA-IVM.
  Interventions: Other: Super-GDF9 supplementation during CAPA-IVM
- Conventional CAPA-IVM (Active Comparator): Group 2: The subject's remaining COCs will be cultured in the CAPA step and the IVM step without the addition of Super-GDF9 during CAPA-IVM.
  Interventions: Other: Conventional CAPA-IVM

INTERVENTIONS:
Other: Super-GDF9 supplementation during CAPA-IVM — Group 1: donated COCs will be exposed to Super-GDF9 at 50 ng/ml in both the CAPACITATION and MATURATION culture steps.
  Arms: Super-GDF9 supplementation during CAPA-IVM
Other: Conventional CAPA-IVM — Group 2: The subject's remaining COCs will be cultured in the CAPA step and the IVM step without the addition of Super-GDF9 during CAPA-IVM.
  Arms: Conventional CAPA-IVM

SUMMARY:
CAPA-IVM (In Vitro Maturation) technology is an assisted reproductive method offering significant benefits in terms of safety and treatment costs, particularly for high-risk patients. These include individuals with ovarian hyperstimulation syndrome (OHSS), venous thrombosis, ovarian torsion, or polycystic ovary syndrome (PCOS). However, while the live birth rate in the CAPA-IVM group (35.2%) is comparable to conventional IVF (43.2%), the number of good-quality embryos and cumulative clinical pregnancy rates remain lower. Improving the CAPA-IVM culture process, particularly through the addition of growth factors found in follicular fluid, has shown promise in enhancing oocyte quality.

Growth differentiation factor 9 (GDF9) and Bone morphogenetic protein 15 (BMP15) play critical roles in follicular development, with their heterodimer structure demonstrating the most positive effects on cumulus-oocyte complexes (COCs). Recent studies have identified a potent variant, super GDF9, which is >1000 times more effective than GDF9 and surpasses cumulin, a heterodimeric growth factor. Super GDF9 enhances cumulus cell expansion and oocyte developmental competence, closely mimicking in vivo maturation.

This study investigates the impact of supplementing super GDF9 during CAPA-IVM culture, aiming to improve outcomes of cumulus-oocyte complexes (COCs) from small follicles and ultimately enhance treatment success.

DETAILED DESCRIPTION:
CAPA-IVM (In Vitro Maturation) technology is an assisted reproductive method offering significant benefits in terms of safety and treatment costs, particularly for high-risk patients. These include individuals with ovarian hyperstimulation syndrome (OHSS), venous thrombosis, ovarian torsion, or polycystic ovary syndrome (PCOS) - who typically present with a high number of antral follicles (constituting nearly 15% of all patients). Although the live birth rate following the first transfer in the CAPA-IVM group is 35.2%, which is not statistically different from the conventional IVF group at 43.2% (risk difference: -8.1%; 95% confidence interval: -16.6% to 0.5%), the number of good-quality embryos per cycle and the cumulative clinical pregnancy rate remain lower than in conventional IVF. Therefore, improving the CAPA-IVM culture process to achieve the optimal number and quality of oocytes is essential.

Concurrently, adding growth factors commonly found in follicular fluid to the culture medium represents a remarkable advancement in improving oocyte quality in CAPA-IVM. Some somatic compartments, such as expansion, metabolism, and apoptosis, are regulated by soluble growth factors, known as oocyte secretion factors (OSFs). Two OSFs, Growth differentiation factor 9 (GDF9) and Bone morphogenetic protein 15 (BMP15), have been identified as critical for follicular development and fertility in various species such as mice, sheep, and humans. During IVM culture, both the immature and mature forms of these factors as well as their homo- and heterodimer structures have been tested. Notably, the heterodimer structure has shown the most positive effects on cumulus-oocyte complexes (COCs) during IVM culture.

Although both growth factors exist in homodimeric forms, recent studies have found that the GDF9 and BMP15 heterodimer can also form a more potent growth factor called cumulin. BMP15 activates latent GDF9 in cumulin, leading to strong signaling in granulosa cells via type I receptors (ALK4/5) and SMAD2/3 transcription factors. Biomedically engineered cumulin has been proposed to noticeably improve embryo outcomes in mouse and porcine models. Recently, a modified version of wild-type GDF9, called super GDF9, has been demonstrated to be >1000 times more potent than GDF9 and 4 times more activity than cumulin in SMAD2/3-responsive transcriptional assays in granulosa cells. Previous research has illustrated that adding super GDF9 to CAPA-IVM media in mice induces gene expression in the ovulatory cascade during CAPA-IVM maturation that closely resembles in vivo maturation. Super GDF9 effectively promotes cumulus cell expansion and enhances oocyte developmental competence in vitro. Hence, super GDF9 can potentially replace cumulin, which faces challenges in production and purification.

This study investigates the impact of supplementing super GDF9 during CAPA-IVM culture, aiming to improve outcomes of cumulus-oocyte complexes (COCs) from small follicles and ultimately enhance treatment success.

This study will recruit 300 COCs (an estimated 10 needed patients). 100 COCs will be allocated to the research arm (sGDF-9), while 200 COCs will be allocated to the control arm.

* Screening for eligibility

  * This study will be conducted at My Duc Hospital, Ho Chi Minh City, Vietnam.
  * Women who are potentially eligible will be provided information about the study at the time of IVM treatment indication.
  * Screening for eligibility will be performed on the day of the first visit when the IVM treatment is indicated.
  * Patients will be provided information about the study and informed consent documents. The investigators will obtain signed informed consent forms from all women before enrollment.
  * Eligible women will be scheduled to undergo oocyte pick-up procedures within 1-7 days from informed consent.
* Oocytes retrieval The oocyte pick-up procedure will be conducted according to the center's standard practices for CAPA-IVM cycles.

Cumulus-oocyte complexes (COCs) from small follicles after OPU will be divided into 2 groups:

* Group 1 (sGDF-9): donated COCs will be cultured in the CAPA and IVM steps, adding 50ng/ml Super-GDF9 during both steps in CAPA-IVM
* Group 2 (Control): The subject's remaining COCs will be cultured in the CAPA and IVM steps without adding Super-GDF9 during CAPA-IVM.

Groups 1 and 2: Collecting after the capacitation step: spent media and blank wells. Collecting after the maturation step: spent media, cumulus cell, and blank wells.

+ CAPA and Maturation culture: CAPA and Maturation culture will be performed routinely following current laboratory protocols. ICSI will be used to fertilize mature oocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 18 and 38 years (both inclusive)
2. BMI ≤ 32 kg/m2
3. PCOS women according to the Rotterdam criteria (2003)
4. Indicating CAPA-IVM treatment.
5. Serum AMH ≥ 4 ng/mL (28.57 pmol/L) at screening and having at least 24 antral follicles in two ovaries by transvaginal ultrasound at the time of CAPA-IVM indication
6. Willing to donate COCs for research purposes
7. Agreeing for frozen embryo
8. Signed informed consent before any study-related procedures

Exclusion Criteria:

1. Known endometrioma or grade 3-4 endometriosis according to ASRM classification
2. Uterine abnormalities
3. Couples with severe male factor (sperm concentration <5 million/ml, motility < 10%), surgical sperm retrieval.
4. Previous history of unexplained immature oocytes after IVF treatment
5. Cycles using donor oocytes

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maturation rate per COC | Two days after oocyte retrieval
  Number of MII / COCs

SECONDARY OUTCOMES:
Maturation rate per patient | Two days after oocyte retrieval
  Number of MII / patient
Degeneration rate per COC | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of degenerated oocytes after IVM / COCs
Degeneration rate per MII | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of degenerated oocytes after IVM / MII
Degeneration rate per patient | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of degenerated oocytes after IVM / patients
t2PN | 16-18 hours after Intra-cytoplasmic sperm injection
  Time of two pronuclei appearance
Fertilization rate per COC | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of fertilized oocytes / COCs
Fertilization rate per MII | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of fertilized oocytes / MII
Fertilization rate per patient | 16-18 hours after Intra-cytoplasmic sperm injection
  Number of fertilized oocytes / patients
Abnormal fertilization rate per COC | 16-18 hours after Intra-cytoplasmic sperm injection
  The percentage of zygotes with 1,3, or more than 3 pronuclei after Intra-cytoplasmic sperm injection / COCs
Abnormal fertilization rate per MII | 16-18 hours after Intra-cytoplasmic sperm injection
  The percentage of zygotes with 1,3, or more than 3 pronuclei after Intra-cytoplasmic sperm injection / MII
Abnormal fertilization rate per patient | 16-18 hours after Intra-cytoplasmic sperm injection
  The percentage of zygotes with 1,3, or more than 3 pronuclei after Intra-cytoplasmic sperm injection / patients
tPNf | 23-25 hours after Intra-cytoplasmic sperm injection
  Time of pronuclei fading
t2 | 25-27 hours after Intra-cytoplasmic sperm injection
  First time frame at which an embryo reaches 2-cell stage blastomeres
t3 | 25-42 hours after Intra-cytoplasmic sperm injection
  First time frame at which an embryo reaches 3-cell stage blastomeres
t4 | 42-44 hours after Intra-cytoplasmic sperm injection
  First time frame at which an embryo reaches 4-cell stage blastomeres
t5 | 44-67 hours after Intra-cytoplasmic sperm injection
  First time frame at which an embryo reaches 5-cell stage blastomeres
t8 | 67-69 hours after Intra-cytoplasmic sperm injection
  First time frame at which an embryo reaches 8-cell stage blastomeres
tSC | During day 3 after intracytoplasmic sperm injection (beginning of the compaction of blastomeres)
  First evidence of compaction
Day-3 embryo rate per COC | Five days after oocyte retrieval
  Counting the number of patients with Day-3 embryo/COCs
Day-3 embryo rate per MII | Three days after Intra-cytoplasmic sperm injection
  Counting the number of patients with Day-3 embryo/ MII
Day-3 embryo rate per patient | Three days after Intra-cytoplasmic sperm injection
  Counting the number of patients with Day-3 embryo / patients
Good quality Day-3 embryos per COC | Three days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 Day-3 embryos / COCs
Good quality Day-3 embryos per MII | Three days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 Day-3 embryos / MII
Good quality Day-3 embryos per patient | Three days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 Day-3 embryos / patients
tM | During day 4 after Intra-cytoplasmic sperm injection
  Time of completion of compaction process
tSB | During day 4 after Intra-cytoplasmic sperm injection (in which the blastocoel is visible)
  Initiation of blastulation
tB | During day 4 after Intra-cytoplasmic sperm injection (before zona starts to thin)
  Full blastocyst
Blastocyst rate per COC (day 5 or 6 embryo) | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of patients with Day-5 or Day-6 embryo/COCs
Blastocyst rate per MII | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of patients with Day-5 or Day-6 embryo/MII
Blastocyst rate per patient | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of patients with Day-5 or Day-6 embryo/patient
Good quality blastocysts per COC | Five or six days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 blastocysts / COCs
Good quality blastocysts per MII | Five or six days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 blastocysts / MII
Good quality blastocysts per patient | Five or six days after Intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 blastocysts / patients
Frozen blastocysts rate per COC | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of frozen blastocysts/ COCs
Frozen blastocysts rate per MII | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of frozen blastocysts/ MII
Frozen blastocysts rate per patient | Five or six days after Intra-cytoplasmic sperm injection
  Counting the number of frozen blastocysts/ patient
The relative expression ratio (R) of human cumulus cell genes | Cumulus cells will be collected and frozen within 30-50 minutes after oocyte denudation, stored at -80oC until RNA purification
  Cumulus cells will be collected, cDNA synthesis after mRNA purification, relative quantification PCR for detecting gene expression (results potentially reported separately)
Rates of Blastocysts by Chromosomal Status in PGT | After study completion, an average of 1 year.
  PGT will be performed to classify blastocysts as euploid, aneuploid or mosaic (results potentially reported separately)
Epigenetic Evaluation | After study completion, an average of 1 year.
  Epigenetic evaluation of blastocysts will be performed by post-bisulfite adaptor tagging (PBAT), and the average DNA-methylation (%) at imprinted germline differentially methylated regions (gDMRs) will be calculated (results potentially reported separately)

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine, the Society of Reproductive Biologists and Technologists, and the Society for Assisted Reproductive Technology. Electronic address: jgoldstein@asrm.org. In vitro maturation: a committee opinion. Fertil Steril. 2021 Feb;115(2):298-304. doi: 10.1016/j.fertnstert.2020.11.018. Epub 2020 Dec 24. PMID 33358333
- [Background] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Smitz J, Gilchrist RB, Norman RJ, Mol BW. In-vitro maturation of oocytes versus conventional IVF in women with infertility and a high antral follicle count: a randomized non-inferiority controlled trial. Hum Reprod. 2020 Nov 1;35(11):2537-2547. doi: 10.1093/humrep/deaa240. PMID 32974672
- [Background] Gilchrist RB, Ho TM, De Vos M, Sanchez F, Romero S, Ledger WL, Anckaert E, Vuong LN, Smitz J. A fresh start for IVM: capacitating the oocyte for development using pre-IVM. Hum Reprod Update. 2024 Jan 3;30(1):3-25. doi: 10.1093/humupd/dmad023. PMID 37639630
- [Background] Herta AC, von Mengden L, Akin N, Billooye K, Coucke W, van Leersum J, Cava-Cami B, Saucedo-Cuevas L, Klamt F, Smitz J, Anckaert E. Characterization of carbohydrate metabolism in in vivo- and in vitro-grown and matured mouse antral folliclesdagger. Biol Reprod. 2022 Oct 11;107(4):998-1013. doi: 10.1093/biolre/ioac124. PMID 35717588
- [Background] Stocker WA, Walton KL, Richani D, Chan KL, Beilby KH, Finger BJ, Green MP, Gilchrist RB, Harrison CA. A variant of human growth differentiation factor-9 that improves oocyte developmental competence. J Biol Chem. 2020 Jun 5;295(23):7981-7991. doi: 10.1074/jbc.RA120.013050. Epub 2020 Apr 29. PMID 32350111
- [Background] Akin N, Ates G, von Mengden L, Herta AC, Meriggioli C, Billooye K, Stocker WA, Ghesquiere B, Harrison CA, Cools W, Klamt F, Massie A, Smitz J, Anckaert E. Effects of lactate, super-GDF9, and low oxygen tension during bi-phasic in vitro maturation on the bioenergetic profiles of mouse cumulus-oocyte complexdagger. Biol Reprod. 2023 Oct 13;109(4):432-449. doi: 10.1093/biolre/ioad085. PMID 37531262
- [Background] Krisher RL, Bavister BD. Enhanced glycolysis after maturation of bovine oocytes in vitro is associated with increased developmental competence. Mol Reprod Dev. 1999 May;53(1):19-26. doi: 10.1002/(SICI)1098-2795(199905)53:13.0.CO;2-U. PMID 10230813
- [Background] Ortmann B, Druker J, Rocha S. Cell cycle progression in response to oxygen levels. Cell Mol Life Sci. 2014 Sep;71(18):3569-82. doi: 10.1007/s00018-014-1645-9. Epub 2014 May 25. PMID 24858415
- [Background] Mottershead DG, Sugimura S, Al-Musawi SL, Li JJ, Richani D, White MA, Martin GA, Trotta AP, Ritter LJ, Shi J, Mueller TD, Harrison CA, Gilchrist RB. Cumulin, an Oocyte-secreted Heterodimer of the Transforming Growth Factor-beta Family, Is a Potent Activator of Granulosa Cells and Improves Oocyte Quality. J Biol Chem. 2015 Sep 25;290(39):24007-20. doi: 10.1074/jbc.M115.671487. Epub 2015 Aug 8. PMID 26254468
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Practice Committee of the American Society for Reproductive Medicine. Endometriosis and infertility: a committee opinion. Fertil Steril. 2012 Sep;98(3):591-8. doi: 10.1016/j.fertnstert.2012.05.031. Epub 2012 Jun 15. PMID 22704630
- [Background] Saenz-de-Juano MD, Ivanova E, Romero S, Lolicato F, Sanchez F, Van Ranst H, Krueger F, Segonds-Pichon A, De Vos M, Andrews S, Smitz J, Kelsey G, Anckaert E. DNA methylation and mRNA expression of imprinted genes in blastocysts derived from an improved in vitro maturation method for oocytes from small antral follicles in polycystic ovary syndrome patients. Hum Reprod. 2019 Sep 29;34(9):1640-1649. doi: 10.1093/humrep/dez121. PMID 31398248
- [Background] Vuong LN, Nguyen MHN, Nguyen NA, Ly TT, Tran VTT, Nguyen NT, Hoang HLT, Le XTH, Pham TD, Smitz JEJ, Mol BW, Norman RJ, Ho TM. Development of children born from IVM versus IVF: 2-year follow-up of a randomized controlled trial. Hum Reprod. 2022 Jul 30;37(8):1871-1879. doi: 10.1093/humrep/deac115. PMID 35595193